CLINICAL TRIAL: NCT05280886
Title: Multi-site Cohort Study for the Development of Personalized Pharmacotherapy in Patients With Tuberculosis (TB)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Inje University (Other)
Collaborators: Ministry of Science and ICT, Republic of Korea (Other Government)
Responsible Party: Principal Investigator, Jae-Gook Shin, Director of Center, Inje University
Other Study IDs: cPMTb-001
Record Dates: First submitted 2022-01-25; First posted 2022-03-15 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Tuberculosis; Latent Tuberculosis; Nontuberculous Mycobacterium Infection
Keywords: TB; Latent Tuberculosis Infection (LTBI); NTM
MeSH Terms: conditions — Tuberculosis; Latent Tuberculosis; Mycobacterium Infections, Nontuberculous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — Whole blood, Plasma, Dried Blood Spot(DBS)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: therapeutic drug monitoring(TDM) — Based on this data, population pharmacokinetic models of antibiotics drugs that can be applicable to TDM will be developed.

SUMMARY:
Based on the collected antibiotic concentration data and individual patient's clinical information, a pharmacokinetic analysis report that can be applied for dose adjustment of the individual patient is provided. The pharmacokinetic/pharmacodynamic index using the minimum inhibition concentration (MIC) of the antibiotic obtained from the patient's clinical isolate is also explored. Utilizing these, we intend to establish a population pharmacokinetic model of antibiotics prescribed in treating Tuberculosis and Nontuberculous mycobacteria (NTM). The developed population pharmacokinetic model can be applied for therapeutic drug monitoring (TDM) based on dose adjustment through the obtained pharmacokinetic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Tuberculosis.
* Latent tuberculosis, or Nontuberculous mycobacteria (NTM) disease and currently under treatment with antibiotic drugs.
* Patients who understand and voluntarily sign an informed consent form before any study-related procedures are conducted.

Exclusion Criteria:

- Children (minors) for whom the consent of a legal representative is impossible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Outpatient and Inpatient who are diagnosed with Tuberculosis, Latent tuberculosis or Nontuberculous mycobacteria (NTM) disease and currently under treatment with antibiotics drugs.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-07-24 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
The maximum plasma concentration (Cmax) | Around 2 weeks or later after the first administration of antibiotics
Area under the plasma concentration versus time curve (AUC) | Around 2 weeks or later after the first administration of antibiotics
Development of population pharmacokinetic (PK) model of antibiotics | Through study completion, an average 3 years
  The population pharmacokinetic properties of anti-TB drugs will be identified by plasma drug concentrations, pharmacogenomics genotypes, or clinical information. Population pharmacokinetic analysis will be performed by using NONMEN Ⅶ software. (ICON development solutions, Ellicott city, Maryland, USA)
AUC/MIC | Through study completion, an average 3 years
  If MIC data is available.
Cmax/MIC | Through study completion, an average 3 years
  If MIC data is available.
Time above MIC (T > MIC) | Through study completion, an average 3 years
  If MIC data is available.

SECONDARY OUTCOMES:
N-acetyltransferase 2(NAT2) Pharmacogenetic analysis | baseline, pre-procedure
  The six single nucleotide polymorphism (SNP) of NAT2, i.e., genotypes: rs1801279 for 191G>A, rs1041983 for 282C>T, rs1801280 341T>C, rs1799930 for 590G>A, rs1208 for 803A>G, and rs1799931 for 857G>A, will be analyzed with SNaPshot® kit (measurement tool) and categorized phenotypes of patients into rapid, intermediate, and slow acetylator.
Solute carrier organic anion transporter family member 1B1(SLCO1B1) Pharmacogenetic analysis | baseline, pre-procedure
  The two SNP of SLCO1B1, i.e., genotypes: rs2306283, rs4149056, will be analyzed with SNaPshot® kit and categorized phenotypes of patients into normal, intermediate, low transporter function.
Biomarker exploration for adverse drug reaction | Through study completion, an average 3 years

CONTACTS AND LOCATIONS:
Overall Officials: JaeGook JaeGook, Study Chair — In-Je University PharmacoGenomics Research Center
Locations (3):
- Indonesia (2):
  - General Hospital Dr. Soetomo, Surabaya, East Java
  - Ibnu Sina Hospital, Gresik, Perum Grand
- Inje University Busan Paik Hoapital Clinical Trial Center, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seo WJ, Koo HK, Kang JY, Kang J, Park SH, Kang HK, Park HK, Lee SS, Choi S, Jang TW, Shin KC, Oh JY, Choi JY, Min J, Choi YK, Shin JG, Cho YS. Risk adjustment model for tuberculosis compared to non-tuberculosis mycobacterium or latent tuberculosis infection: Center for Personalized Precision Medicine of Tuberculosis (cPMTb) cohort database. BMC Pulm Med. 2023 Nov 24;23(1):471. doi: 10.1186/s12890-023-02646-7. PMID 38001469
- [Derived] Soedarsono S, Jayanti RP, Mertaniasih NM, Kusmiati T, Permatasari A, Indrawanto DW, Charisma AN, Lius EE, Yuliwulandari R, Quang Hoa P, Ky Phat N, Thu VTA, Ky Anh N, Ahn S, Phuoc Long N, Cho YS, Shin JG. Development of population pharmacokinetics model and Bayesian estimation of rifampicin exposure in Indonesian patients with tuberculosis. Tuberculosis (Edinb). 2023 Mar;139:102325. doi: 10.1016/j.tube.2023.102325. Epub 2023 Feb 14. PMID 36841141